CLINICAL TRIAL: NCT02351843
Title: Efficacy and Safety of Low Amplitude Electroconvulsive Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Device Feasibility
Other Study IDs: Pro00058639
Record Dates: First submitted 2015-01-27; First posted 2015-01-30 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2016-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 500 mA ECT (Experimental): Right unilateral, ultra brief pulse ECT, with 500 mA current amplitude
  Interventions: Device: MECTA Spectrum 5000Q
- 800 mA ECT (Active Comparator): Right unilateral, ultra brief pulse ECT, with 800 mA current amplitude
  Interventions: Device: MECTA Spectrum 5000Q

INTERVENTIONS:
Device: MECTA Spectrum 5000Q

SUMMARY:
The purpose of this study is to demonstrate the clinical feasibility of low amplitude electroconvulsive therapy (ECT) to reduce, and possibly eliminate the side effects of ECT by lowering the strength of the ECT stimulus from the conventional 800 mA to 500 mA. Low amplitude ECT could potentially reduce the risks associated with ECT while preserving its unparalleled efficacy. This novel development would remove key obstacles to allow for the wider adoption of ECT as a safe and effective therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, age 18-70
2. DSM-IV-TR diagnosis of major depressive episode in unipolar or bipolar disorder, confirmed by the MINI-PLUS
3. MMSE total score > 26
4. Referred for ECT
5. Competent to provide informed consent
6. Able to read or comprehend English

Exclusion Criteria:

1. Lifetime history of schizophrenia, schizoaffective disorder, mental retardation
2. Current neurostimulation treatment (e.g., ECT, magnetic seizure therapy, transcranial magnetic stimulation, vagus nerve stimulation, deep brain stimulation)
3. Current alcohol abuse or dependence within past 6 months
4. Current substance abuse or dependence within past 6 months
5. History of central nervous system (CNS) disease
6. Current diagnosis of dementia or delirium
7. MoCA total score < 26
8. Current visual, auditory, or motor impairment that compromises ability to complete evaluations
9. Patients with intracranial implants
10. MRI contraindications: pregnancy, implanted metal, and claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in California Verbal Learning Test-II | Baseline and within 24 to 48 hours of each ECT session

OTHER OUTCOMES:
Change in Hamilton Rating Scale for Depression 24-item | Baseline and within 24 to 48 hours of each ECT session
Change in Quick Inventory of Depressive Symptomatology Clinician Rated and Self Report | Baseline and within 24 to 48 hours of each ECT session
Change in Brief Visuospatial Memory Test-Revised | Baseline and within 24 to 48 hours of each ECT session
Change in Autobiographical Memory Interview Test | Baseline and within 24 to 48 hours of each ECT session
Change in Delis Kaplan Executive Function System | Baseline and within 24 to 48 hours of each ECT session
Change in Trail Making Test Part A | Baseline and within 24 to 48 hours of each ECT session
Change in Grooved Pegboard test | Baseline and within 24 to 48 hours of each ECT session

CONTACTS AND LOCATIONS:
Locations (1):
- DukeUMC, Durham, North Carolina, United States